CLINICAL TRIAL: NCT04336709
Title: Comparison of Anti-microbial Efficacy of Calcipex and Metapex in Endodontic Treatment of Chronic Apical Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Momina Anis Motiwala, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-0304-3229
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Chronic Apical Periodontitis
Keywords: intracanal medicament; medicament removal; bacterial culture; efficacy; oil based medicament; colony forming unit
MeSH Terms: interventions — calcipex II; Metapex

STUDY DESIGN:
Intervention Model Description: First visit: After chemomechanical preparation, irrigation and drying, a sterile paper point (size 20; EZ Endo, USA) will be inserted to the confirmed working length of the canal, and retained in position for 60 seconds for sampling (S1). Afterwards, the paperpoint will be gently removed and placed in an eppendorf tube (5 ml) containing Brain Heart Infusion Broth and sent directly to the microbiology laboratory for microbial cultivation. Respective intracanal medicament will be placed by means of lentulo spiral fillers and packed with a cotton pellet at the level of canal entrance. Access cavity will be filled with a temporary filling, Cavit-G. Second visit after 7 day, medicament will be removed. In case of Metapex (oil based medicament) either Protaper rotary or ultrasonic activation of file will be used for removal and radiograph obtained to ensure removal and sample will be obtained(S2). The canals will be then obturated. A definitive restoration will be placed subsequently.
Who Masked: Investigator, Outcomes Assessor
Masking Description: the participant or the care provider cannot be masked due to difference in colors of the medicaments, Metapex being yellow. The investigator (lab technician) and outcome assessor will be masked regarding the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcipex II (Active Comparator): Calcipex group Manufactures Nishika, Yamaguchi, Japan Color- White Formulation- Water based Duration- 7 days Form: Paste Frequency: Used once on 1st day only till canal fills. Composition- Water-based calcium hydroxide paste without radio contrast agent (Barium Sulfate) Packaging- (1 syringe of Calcipex Plain II (1.8g), 2 needles of Nishika Spin with 2 needle caps) Storage requirement- Room temperature (1-30℃).
  Interventions: Drug: Calcipex II
- Metapex (Active Comparator): Metapex group Manufactures- Meta Biomed, Korea Color- Yellow Formulation- Oil based Duration- 7 days Form: Paste Frequency: Used once on 1st day only till canal fills. Composition- Premixed oil-based paste composed of Calcium Hydroxide with Iodoform and silicon oil Packaging-2.2g paste in 1 syringe. 20 disposable tips. 1 ring rotator for direction control of the tip Storage requirement- Room temperature (1-30℃).
  Interventions: Drug: Metapex

INTERVENTIONS:
Drug: Calcipex II — Water based intracanal medicament
  Arms: Calcipex II
Drug: Metapex — Oil based intracanal medicament
  Arms: Metapex

SUMMARY:
Introduction:

Pulpal necrosis may lead to spread of the infection from the pulp to involve the apex of the tooth and surrounding bone which when asymptomatic with periapical radiolucency on radiograph, is called chronic apical periodontitis. In order to eliminate the virulent bacteria and to overcome the inflammation in the root apex, endodontic treatment is the treatment of choice. Bacteria usually survive in the complex anatomy of the root canal system. In order to eliminate the remaining bacteria, various intracanal medicaments have been used widely however, there is controversy over their use and efficacy. Calcium hydroxide (CH) is the most commonly used intracanal medicament between root canal treatment sessions and available in different combinations. Multiple studies have been conducted to evaluate the effect of various types of CH based medicaments but whether CH with iodoform is more effective than CH alone against endodontic pathogens is a matter of controversy. In order to evaluate the true reduction in microbial load from the infected canals, microbial culture is a predictable and convenient tool.

Thus, this study aims to evaluate the antimicrobial effectiveness of inter-appointment intracanal medicament with either CH alone (Calcipex) or CH with iodoform (Metapex) for the treatment of infected root canals of teeth diagnosed with chronic apical periodontitis using colony forming unit (CFU).

Objective: To compare the anti-microbial efficacy of calcipex and metapex in endodontic treatment of teeth diagnosed with chronic apical periodontitis and to compare two different methods for removal of oil based intracanal medicaments.

Method: Approval from ERC is obtained. The selected subjects will be divided in to two study groups using a computer generated randomization list i.e., Group A - Calcipex group (n = 30) and Group B - Metapex group (n = 30). Two samples will be collected from the root canals for evaluation of microbial load after chemomechanical preparation (S1) (before use of intracanal medicament) and after usage of intra canal medicament (S2)(after 7 days).

Two techniques will be used for removal of oil based medicaments. Two radiographs will be obtained for each technique, after oil based medicament placement and after medicament removal for evaluation.

Data Analysis: Mean and standard deviation of continuous variable will be computed. Frequency distribution and proportion of categorical variables will be determined. Paired t-test will be used to assess difference bet¬ween antimicrobial efficacies within groups of medicaments. Independent sample t-test will be used to assess antimicrobial efficacies between groups. Level of significance will be kept at 0.05.

Mann whitney U test will be used to evaluate medicament removal between 2 groups and at three canal levels; coronal, middle and apical.

DETAILED DESCRIPTION:
This study aims to evaluate the antimicrobial effectiveness of inter-appointment intracanal medicament with either CH alone (Calcipex) or CH with iodoform (Metapex) for the treatment of infected root canals of teeth diagnosed with chronic apical periodontitis.

And, to compare the effectiveness of rotary master apical file with ultrasonic activation of endodontic file in the removal of oil based intracanal medicament from the canal.

Risk / Benefit Assessment At this point investigators are not anticipating any risk related to the trial intervention.

TRIAL DESIGN: Two-arm parallel design, Randomized controlled trial. SETTING: Dental Clinics, Aga Khan University Hospital, Karachi

EXPECTED DURATION OF TRIAL:

Study Duration: Four months after registration By visit: 2 visits, with followup period of 7 days±3 after the first visit.

CRITERIA FOR EVALUATION Primary Efficacy Endpoint Reduction in microbial load (CFU/ml) at 7 days after use of intracanal medicament Safety Evaluations No Incidence of adverse events with any agent

Investigational product management: The investigator will purchase the drug locally and will label and store in safe and secure place. The product can be stored at room temperature i.e.1-30℃

Sampling technique: Non probability purposive sampling Sampling size: Sample size was calculated using WHO sample size calculator. Dutta et al.16 showed that the population mean and SD of teeth treated with calcium hydroxide based intracanal medicaments were 50.3±13 CFU/mL. Keeping the absolute precision at 0.05 and level of confidence at 95%, the required sample size turned out to be 26 teeth. The sample is inflated to 30. As tthere are two groups, therefore, a total of 60 teeth will be taken.

RANDOMIZATION, BLINDING AND TREATMENT ALLOCATION:

The selected subjects will be assigned to one of the two study groups only known to the researcher who is not involved in the outcome assessment using block randomization. This would be facilitated by CTU. The block size would be 6.

Group A (Control group) - Calcipex group (n = 30) Group B (Intervention group) - Metapex group (n = 30) The sample in eppendorff tubes will be sent in a zip lock bag to the microbiology laboratory labeled with either group A or B. Patient, analyzer and the statistician will be blinded about the intervention groups. The recruitment of patients, collection of samples and placement of intracanal medicament will be performed by a single investigator.

POSSIBLE RISKS OR BENEFITS:

There is no risk involved in this study as the study is based on routine procedure of endodontic treatment. It will be a benefit for future patients which will help us to decide which intracanal medicament is more effective to use in infected canals.

DATA COLLECTION INSTRUMENTS The data will be collected on case report form (CRF) on first and second visit. The CRF has been developed by investigator and reviewed by experts of the field. Data will be stored in a password protected database. To assure quality, data will be double checked to avoid discrepancies and errors.

PATIENT CONFIDENTIALITY, ACCESS AND STORAGE:

The information provided by the participant will remain confidential. Nobody except investigators will have access to it. Participants' name and identity will not be disclosed at any time. However, the data may be seen by ethical review committee, DSMB or any local regulatory body. As per GCP and other guidelines, data will be retained for 3 years.

ETHICAL CONSIDERATIONS:

The study will be started after obtaining approval from Institutional Ethics Review Committee(approved already). Patients who fulfilled the inclusion criteria will receive detailed information regarding the study and only those participants will be recruited who will sign the written consent form. The study will be conducted according to the World Medical Association's Declaration of Helsinki and the principles of GCP (Good Clinical Practice). Any subsequent protocol amendments will be submitted to ERC and regulatory authorities for approval. The trial will be conducted in compliance with regulations, particularly specifying pharmaco-vigilance reporting and a copy of final study report will be submitted to ERC.

DATA COLLECTION PROCEDURE:

First visit: The tooth diagnosed with chronic apical periodontitis will be anesthetized using 2% lidocaine (with 1:100,000 epinephrine) and isolated with the rubber dam. Access opening will be performed using high and low speed round bur. Coronal and radicular necrotic pulp will be extirpated using barbed broaches. The root canal will be initially prepared by using hand K-files (Endoflex; K-File, Size 8-20, NiTi) with quarter turn and pull motion. A 23-gauge side vented needle will be used to deliver 1 mL of sodium hypochlorite for irrigation after each instrument size. The working length will be established with an apex locator and confirmed by the periapical radiographs. Chemo-mechanical preparation will be completed using Protaper Next (Dentsply; Sirona, USA) depending on both root anatomy and initial diameter of the root canal. The preparation will be completed in the same appointment in all cases. After completion of the preparation, the canals will be irrigated with saline and dried with paper points. A sterile paper point (size 20; EZ Endo, USA) will be inserted to the confirmed working length of the canal, and retained in position for 60 seconds for sampling (S1). Afterwards, the paperpoint will be gently removed and placed in an eppendorf tube (5 ml) containing Brain Heart Infusion Broth and sent directly to the microbiology laboratory for microbial cultivation.

In Group A, the canal will be medicated with Calcipex (Calcipex®II, Nishika, Yamaguchi, Japan) which will be placed by means of lentulo spiral fillers and packed with a cotton pellet at the level of canal entrance. Access cavity will be filled with a temporary filling, Cavit-G (3M-ESPE, USA). In Group B, the canal will be medicated with Metapex (Meta Biomed, Korea) using the same protocol as mentioned above.

Second visit: Patient will be followed up on seven +/- 3 days, the tooth will be isolated and the protocol will be followed the same way as described before. The temporary filling will be removed and the paste carried out of the canal by using sterile file and irrigated with normal saline to wash out the medicament. A post medication sample will be taken with the help of sterile paper point in both groups as described previously (S2). The canals will be then obturated with gutta-percha and calcium hydroxide sealer (Sealapex, Kerr Dental, USA) by lateral compaction technique. A definitive restoration will be placed subsequently.

Outcome assessment: It will be done in the microbiology laboratory on the basis of CFU/ml.

RIGHT OF REFUSAL TO PARTICIPATE AND WITHDRAWAL:

Participants will be given choice to either participate or refuse to participate in the study

INCENTIVE:

No incentive will be given to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Single rooted human permanent teeth
* Single root canal clinically diagnosed with chronic apical periodontitis
* No history of antibiotics use in last 3 months.

Exclusion Criteria:

* Periodontally compromised teeth with Grade III mobility.
* Endodontically non-salvageable teeth.
* Immuno-compromised patients/systemic illness.
* Excessive root resorption.
* History of allergy to calcium hydroxide or iodoform.
* Endodontic retreatment cases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Antimicrobial efficacy | 7 days
  antimicrobial efficacy of intracanal medicament as measuring using Colony forming unit/ml via bacterial culture. The higher CFU/ml suggests more bacterial colonies. We expect the counts to reduce after using the intracanal medicament

SECONDARY OUTCOMES:
Efficacy of intracanal medicament removal | 7 days
  Efficacy of intracanal medicament removal using four grade scoring system given by Khademi et al to evaluate amount of medicament remnant in the canal as seen and evaluated using periapical radiographs.
  GRADING:
  Removal efficacy 0 = the surface was not covered with calcium hydroxide
  1. = 1/3 of the surface was covered with calcium hydroxide
  2. = 2/3 of the surface was covered with calcium hydroxide
  3. = the surface was covered with calcium hydroxide completely Grade 0 and 1 will be taken as effective cleaning Grade 2 and 3 will be taken as non-effective cleaning

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Everything will be managed and reported and collected and available for sharing to remove bias and ensure accurate conductance of study according to given protocols.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 4 months, as soon as we go by the steps till completion of study

REFERENCES:
- [Background] Mozayeni MA, Haeri A, Dianat O, Jafari AR. Antimicrobial effects of four intracanal medicaments on enterococcus faecalis: an in vitro study. Iran Endod J. 2014 Summer;9(3):195-8. Epub 2014 Jul 5. PMID 25031593
- [Background] Martinho FC, Gomes BP. Quantification of endotoxins and cultivable bacteria in root canal infection before and after chemomechanical preparation with 2.5% sodium hypochlorite. J Endod. 2008 Mar;34(3):268-72. doi: 10.1016/j.joen.2007.11.015. Epub 2008 Jan 31. PMID 18291273
- [Background] Manzur A, Gonzalez AM, Pozos A, Silva-Herzog D, Friedman S. Bacterial quantification in teeth with apical periodontitis related to instrumentation and different intracanal medications: a randomized clinical trial. J Endod. 2007 Feb;33(2):114-8. doi: 10.1016/j.joen.2006.11.003. PMID 17258626
- [Background] Gautam S, Rajkumar B, Landge SP, Dubey S, Nehete P, Boruah LC. Antimicrobial efficacy of metapex (calcium hydroxide with iodoform formulation) at different concentrations against selected microorganisms--an in vitro study. Nepal Med Coll J. 2011 Dec;13(4):297-300. PMID 23016485
- [Derived] Motiwala MA, Habib S, Ghafoor R, Irfan S. Comparison of antimicrobial efficacy of Calcipex and Metapex in endodontic treatment of chronic apical periodontitis: a randomised controlled trial study protocol. BMJ Open. 2021 Jul 21;11(7):e048947. doi: 10.1136/bmjopen-2021-048947. PMID 34290069